CLINICAL TRIAL: NCT03188731
Title: Pregnant Women (PW) Cohort for Evaluation of Risks of Congenital Malformations and Other Adverse Pregnancy Outcomes After Zika Virus Infection (Part of ZIKAlliance)
Brief Title: ZIKAlliance Pregnant Women Cohort
Acronym: ZIKAlliancePW
Status: Completed | Type: Observational
Sponsor: University of Heidelberg Medical Center (Other)
Collaborators: European Union (Other); ZIKAlliance (Unknown); Oswaldo Cruz Foundation (Other); University of Sao Paulo (Other); London School of Hygiene and Tropical Medicine (Other); Federal University of Bahia (Other); Universidade Federal de Goias (Other); University Medical Center Groningen (Other); University of Carabobo (Other); Universidad Industrial de Santander (Other); Sosecali Hospital, Guyaquil (Unknown); Instituto de Medicina Tropical "Pedro Kourí (IPK), Cuba (Unknown); Mexican National Institute of Public Health (Other Government); Instituto Mexicano del Seguro Social (Other Government); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Thomas Jaenisch, Senior Scientist, University of Heidelberg Medical Center
Other Study IDs: 734548PW (EC | H2020 | RIA)
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Zika Virus; Pregnancy Related
Keywords: ZIKA; Dengue; Chikungunya; Pregnant Women; Pregnant Woman; ZIKV
MeSH Terms: conditions — Zika Virus Infection; Dengue; Chikungunya Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Hair, Urine, Vaginal fluids, Saliva, Semen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant Women

SUMMARY:
The aim of this proposal is to evaluate the causal relationship between Zika virus (ZIKV) infections in pregnancy and congenital malformations. We will estimate the absolute and relative risks of congenital malformations and other adverse outcomes of pregnancy among women who become infected with ZIKV during pregnancy compared to uninfected pregnant women, also leading to further validation of the Congenital Zika Syndrome.

DETAILED DESCRIPTION:
The aim of this proposal is to evaluate the causal relationship between Zika virus (ZIKV) infections in pregnancy and congenital malformations. We will estimate the absolute and relative risks of congenital malformations and other adverse outcomes of pregnancy among women who become infected with ZIKV during pregnancy compared to uninfected pregnant women, also leading to further validation of the Congenital Zika Syndrome.

We will also determine the ZIKV maternal to child transmission rate and evaluate co-factors or effect modifiers that account for the large variability seen in the preliminary absolute risk estimates derived from population figures and reporting of microcephaly in different states in Brazil and across Latin America.

We will carry out a pregnant women (PW) multicentre cohort study in areas across Latin America and the Caribbean. Women will be enrolled early in pregnancy and followed every 4 weeks, in connection with their routine antenatal care visits. At each visit, urine and blood samples will be collected, tested and stored.

Among PW reporting recent or current undifferentiated fever/rash syndrome at any point in time, the acute illness episode will be characterized in greater detail. PW with suspected ZIKV infection (i.e. meeting the Pan American Health Organization (PAHO) clinical case definition) during pregnancy will be managed according to national protocols. Irrespective of symptoms, pregnant women will be followed prospectively and revisited at birth (or after abortion) for a detailed documentation of the outcome of their pregnancy.

Live newborns will receive a detailed neonatal examination. In the course of examination of the newborns, biological samples will be collected and stored. Other potential causes of congenital abnormalities (TORCHS infections in the mother, toxic substances, chromosomal abnormalities), and potential effect modifiers (for example past flavivirus infections/vaccinations, socio-economic status) will also be assessed.

With appropriate counselling and consent, biological samples of newborns with severe abnormalities, deceased newborns, stillborn babies, and aborted foetuses from ZIKV-infected mothers will be collected to help elucidate the aetiological contribution of ZIKV in neurological and other congenital malformations.

Children of women infected with ZIKV during pregnancy - and a subset of the children born to uninfected women - will be followed prospectively after birth for the assessment of neuro-developmental milestones (separate protocol).

ELIGIBILITY:
Inclusion Criteria:

* at least 16 years old
* Pregnancy status confirmed
* Within first or second trimester or first month of marked transmission season

Exclusion Criteria:

* Planing to leave area
* Unable to attend follow-up visits
* Unable to undergo venipuncture
* Participates in another pregnant women study for ZIKA
* Unable to consent without legal guardian

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Pregnant
Study Population: Pregnant Women
Sampling Method: Probability Sample
Enrollment: 3852 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Congenital Abnormalities | At birth

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Jänisch, Principal Investigator — University Hospital Heidelberg
Locations (14):
- Bolivia (2):
  - Sosecali Ltd. (SOSE), Guaqui
  - INSERM, Santa Cruz
- Brazil (6):
  - Federal University of Bahia (UFB), Bahia
  - Universidade Federal de Minas Gerais, Belo Horizonte
  - Federal University of Goias, Goiás
  - Fundacao Oswaldo Cruz (FIOCRUZ), Recife
  - Fundacao Oswaldo Cruz (FIOCRUZ), Rio de Janeiro
  - University of Sao Paulo, São Paulo
- Industrial University of Santander (UIS), Bucaramanga, Colombia
- Pedro Kouri Institute (IPK), Havana, Cuba
- INSERM, Pointe-à-Pitre, Guadeloupe
- Mexico (2):
  - IMSS Mexico (IMSS), Guadalajara
  - National Institute of Public Health (INSP), Mérida
- Universidad de Carabobo / UMC Groningen (UMCG), Valencia, Venezuela

IPD SHARING:
Plan to Share IPD: Yes
1. The ZIKAlliance birth cohort is part of the 3 EC-funded Zika consortia. The data are intended to be shared after the individual cohort data is analyzed and published.
  2. The ZIKAlliance birth cohort is part of the WHO-moderated IPD meta-analysis Consortium. The data are intended to be shared after the individual cohort data is analyzed and published.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Avelino-Silva VI, Mayaud P, Tami A, Miranda MC, Rosenberger KD, Alexander N, Nacul L, Segurado A, Pohl M, Bethencourt S, Villar LA, Viana IFT, Rabello R, Soria C, Salgado SP, Gotuzzo E, Guzman MG, Martinez PA, Lopez-Gatell H, Hegewisch-Taylor J, Borja-Aburto VH, Gonzalez C, Netto EM, Saba Villarroel PM, Hoen B, Brasil P, Marques ETA, Rockx B, Koopmans M, de Lamballerie X, Jaenisch T; ZIKAlliance Clinical Study Group. Study protocol for the multicentre cohorts of Zika virus infection in pregnant women, infants, and acute clinical cases in Latin America and the Caribbean: the ZIKAlliance consortium. BMC Infect Dis. 2019 Dec 26;19(1):1081. doi: 10.1186/s12879-019-4685-9. PMID 31878895